CLINICAL TRIAL: NCT07117825
Title: Aortic Dissection fAlse enlarGement radIomics predictiOn
Acronym: ADAGIO
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, TINELLI GIOVANNI, Prof, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6518
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Dissection; Aortic Diseases; Aortic Dissection
MeSH Terms: conditions — Aortic Diseases; Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: AORTIC DISSECTION CT SCAN ANALYSIS — Patients with type A or type B acute aortic dissection, treated either with medical therapy or with endovascular/open surgery in the study period and who underwent subsequent radiological follow-up.

SUMMARY:
The objective of this study is to find, in acute phase of aortic dissection, CT scans characteristics through radiomics features, that can help us to predict a significant growth of dissected descending aorta or a false lumen enlargement in order to treat the patient promptly.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previous acute aortic (type A or B) dissection, undergoing medical or surgical therapy and in clinical-radiological follow-up.

Exclusion Criteria:

* Patients with no appropriate radiological follow up;
* Patients who died in the acute phase of aortic type A or B dissection.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with type A or type B acute aortic dissection, treated either with medical therapy or with endovascular/open surgery in the study period and who underwent subsequent radiological follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Predict the false lumen enlargement (>5.5 mm aortic diameter growth at CT follow-up control) through radiomics analysis applied on CT scans. | 24 MONTHS

CONTACTS AND LOCATIONS:
Locations (1):
- Giovanni Tinelli, Roma, Italy

IPD SHARING:
Plan to Share IPD: No